CLINICAL TRIAL: NCT03308578
Title: Statins and CPAP in Adipose Tissue: A Randomized Clinical Trial in Obstructive Sleep Apnea
Brief Title: Statins and CPAP in Adipose Tissue of OSA
Acronym: SCAT-OSA
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Virend Somers, MD, PhD, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 17-005119; R01HL065176 (NIH)
Record Dates: First submitted 2017-10-09; First posted 2017-10-12 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Sleep Apnea, Obstructive
Keywords: Obstructive sleep apnea; Adipose tissue
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Atorvastatin (Experimental): Subjects randomized to this arm will be started on a lower dose of atorvastatin 40 mg daily for the first 4 weeks. If they are tolerating this dose without significant problems, atorvastatin will be increased to 80 mg daily.
  Interventions: Drug: Atorvastatin
- Placebo Oral Capsule (Placebo Comparator): Subjects randomized to this arm will receive placebo capsules matching study drug.
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Atorvastatin — Subjects randomized to this arm will receive 40 mg capsules, once daily dose for the first 4 weeks followed by 2X40mg capsules, once daily dose for remaining 5 months of the study
  Arms: Atorvastatin
Drug: Placebo oral capsule — Subjects randomized to this arm will receive placebo capsules, once daily dose for the first 4 weeks followed by 2X40mg capsules, once daily dose for remaining 5 months of the study
  Arms: Placebo Oral Capsule

SUMMARY:
This study is aimed at examining the alterations in adipose tissue in obstructive sleep apnea (OSA) patients in response to treatment with atorvastatin in continuation with standard treatment with continuous positive airway pressure (CPAP).

DETAILED DESCRIPTION:
In recent years the role adipose tissue to the development of cardiometabolic disorders has been increasingly recognized. Dysfunctional adipose tissue is an important source for systemic inflammation, AngII, and FFA, thus increasing CV risk in obese and aging populations. Even though heightened cardiovascular risk in OSA patients is acknowledged, adipose tissue from OSA patients has not been investigated.

CPAP is standard therapy for OSA, but has shown mixed results for improvement of vascular function, insulin sensitivity, and BP, and does not reduce CV events and mortality, even in patients with established CV disease. Hence, eliminating IH alone may not be sufficient to repair preexisting damage; additional adjunct strategies aimed at cellular repair may be required to reduce cardiometabolic burden and CV risk. Statins have pleiotropic effects including reducing inflammation, and improving BP. The aim of this study is to examine the longitudinal changes in the cellular and molecular composition of adipose tissue in OSA subjects in response to 6 months combination therapy of CPAP and atorvastatin. We hypothesize that the combination therapy will reduce adipose tissue cellular damage (p16INK4A+γ-H2AX dual positive cells). Also, decreases in adipose tissue cellular damage will be associated with improved cardiometabolic profile. These studies will provide pivotal insights into potential therapeutic strategies which may reduce cardiometabolic burden in OSA population.

ELIGIBILITY:
Inclusion Criteria

* Participated in IRB 17-003825
* Apnea hypopnea index, AHI/RDI ≥10, or AHI/RDI >5 with significant nocturnal hypoxemia documented by a fall in oxygen saturation to 90% or below.
* Women of child-bearing age will be allowed to participate if they agree to use acceptable birth control during the study period.
* TSH levels in range of 0.3-6 mIU/L (TSH above 6 mIU/L will be allowed if free thyroxine (free T4) is within normal range)

Exclusion Criteria

* Elevated ALT (>3 times upper normal limit)
* Fasting glucose >120 mg/dL and/or HbA1c ≥ 6.5 %
* Females planning to be pregnant in next six months will not be included in the study
* Known serious or hypersensitivity to HMG-CoA reductase inhibitors.
* Alcohol consumption >3 units/day

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2023-12-12 (Actual); Study Completion 2023-12-12 (Actual)

PRIMARY OUTCOMES:
Changes in prevalence of dual positive p16IND4A and gamma H2AX cells in adipose tissue | Approximately 6 months
  Positivity for both (p16^IND4A and γH2AX) serves as a marker of cellular damage. Fat biopsy from the will be performed to obtain up to 1 gm of adipose tissue. These fat samples will be batched for analysis to determine the prevalence of cellular damage. Biopsy will be obtained at 3 months and 6 month follow-up.

SECONDARY OUTCOMES:
Changes in prevalence of phosphorylated p53 (pp53) in adipose tissue | approximately 6months
  Presence of pp53 as a ratio of phospho to total p53 to access cellular damage in adipose tissue at 3 month and 6 month follow-up
Changes in 24- h mean arterial pressure | approximately 6months
  Changes in ambulatory measure of blood pressure at 3 month and 6 month.
Changes in vascular endothelial function | approximately 6months
  Comparison of change in brachial artery diameter in response to hyperemia at 3 month and 6 month follow-up.
Changes in insulin sensitivity | approximately 6months
  Changes in the measure for area under the curve for glucose and insulin as determined during oral glucose tolerance test at 3 month and 6 month.
Changes in body composition | approximately 6months
  Changes in percentage body fat content at 3 month and 6 month.

CONTACTS AND LOCATIONS:
Overall Officials: Virend Somers, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Bock JM, Vungarala S, Sompalli S, Covassin N, Bukartyk J, Karim S, Louis ES, Wright RS, Singh P, Somers VK. High-Intensity Atorvastatin and 24-Hour Blood Pressure in Obstructive Sleep Apnea: A Randomized, Double-Blind, Placebo-Controlled Pilot Study. Am J Hypertens. 2025 Oct 10:hpaf202. doi: 10.1093/ajh/hpaf202. Online ahead of print. PMID 41072928
- [Derived] Greenlund IM, Bock JM, Govindan N, Kantas D, Singh P, Covassin N, Somers VK. Blood Pressure and Heart Rate Response to Orthostasis in Somali Americans. J Racial Ethn Health Disparities. 2025 Mar 15:10.1007/s40615-025-02389-7. doi: 10.1007/s40615-025-02389-7. Online ahead of print. PMID 40088388
- [Derived] Greenlund I, Bock J, Govindan N, Kantas D, Singh P, Covassin N, Somers V. Blood Pressure and Heart Rate Response to Orthostasis in Somali Americans. Res Sq [Preprint]. 2024 Oct 21:rs.3.rs-4925722. doi: 10.21203/rs.3.rs-4925722/v1. PMID 39502777